CLINICAL TRIAL: NCT04060472
Title: Single-center, Single-arm and Phase II/III Clinical Study of Paclitaxel (Albumin-binding) Combined With Oxaliplatin as First-line Treatment for Advanced Hepatobiliary and Malignant Tumors
Brief Title: Paclitaxel (Albumin-bound) and Oxaliplatin for Advanced Hepatobiliary and Malignant Tumors
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dong Wang (Other)
Responsible Party: Sponsor-Investigator, Dong Wang, Single-center, Single-arm and Phase II/III Clinical Study of Paclitaxel (Albumin-binding) Combined With Oxaliplatin as First-line Treatment for Advanced Hepatobiliary and Malignant Tumors, Third Military Medical University
Organization: Third Military Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ThirdMMUb
Record Dates: First submitted 2019-08-15; First posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Advanced Hepatobiliary and Malignant Tumors
MeSH Terms: conditions — Neoplasms | interventions — Albumin-Bound Paclitaxel; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- albumin-bound paclitaxel + oxaliplatin (Experimental)
  Interventions: Drug: albumin-bound paclitaxel + oxaliplatin

INTERVENTIONS:
Drug: albumin-bound paclitaxel + oxaliplatin — Using albumin-bound paclitaxel (125 mg/m2, d1, 8, 15, ivgtt) + oxaliplatin (80 mg/m2, d1, 8, ivgtt) with or without other chemotherapeutic drugs, 28 days /cycle, until the disease progresses or patients can not tolerate toxicity. The investigators decide the follow-up treatment plan.

SUMMARY:
1. Advantages of albumin-bound paclitaxel Paclitaxel for injection (albumin-binding type) uses human serum albumin (HAS) as a carrier, and paclitaxel and HSA are made into paclitaxel-bound albumin nanoparticles by a high-pressure homogenization technique. After injection of paclitaxel (albumin-binding) into the blood, it rapidly disintegrates and disperses into a smaller albumin-paclitaxel complex, which binds and activates the gp60 albumin receptor on vascular endothelial cells, interacts with Caveolin on the cell membrane, and then is transported to the tumor intercellular substance by transcytosis. Tumor cells can secrete a SPARC protein with a specific affinity for albumin, which actively captures the albumin-paclitaxel complex in the tumor stroma and accumulates around the tumor cells. Since tumor neovascular endothelial cells highly express gp60 receptor and the SPARC protein is also highly expressed in the tumor region, the special transport mechanism of "gp60- Caveolin / caveola -SPARC protein" makes the paclitaxel for injection (albumin binding) have unique targeting and penetrating properties toward tumor tissues, hence the drug is highly concentrated in the tumor tissue, which can better increase the therapeutic effect and reduce the damage to normal tissues.

Paclitaxel for injection (albumin-binding type) has the following advantages: (1) it is unnecessary to pre-administer anti-allergic drugs, the infusion time is within 30 min, and patients have good compliance; (2) due to its higher safety, the dosage can be given as high as 260-300 mg/m2; (3) it makes full use of gp60 / cysteine acid secretory protein (SPARC protein) channel to make the drug enrich toward the tumor area, and the effect is good; (4) as the dosage is within 80 ~ 300 mg/m2, the AUC increase proportionally with the administered dose, ]the body is linearly metabolized., the half-life period does not prolong with the dose, and the clinical medication is safe and controllable. Currently, the drug has been approved for breast cancer treatment in China; approved by the US Food and Drug Administration (FDA) for breast cancer, lung cancer, and pancreatic cancer treatment; approved for gastric cancer treatment in Japan; and NCCN guidelines recommend it for the treatment of intrahepatic cholangiocarcinoma, melanoma, ovarian cancer, and cervical cancer.

In summary, based on the biological advantages of albumin-binding paclitaxel such as high-distribution, high-dose, high-efficiency, and low-toxicity, the reported good clinical benefit and safety for hepatobiliary and malignant tumors, and the limited data about albumin-bound paclitaxel + oxaliplatin as the first-line treatment for advanced hepatobiliary and pancreatic malignancies, especially in Chinese patients, our center believes that is feasible and necessary to explore the effectiveness and safety of paclitaxel for injection (albumin-binding) combined with oxaliplatin as the first-line drugs for treatment of advanced oxaliplatin-based malignant tumors.

2 Purposes To evaluate the efficacy and safety of paclitaxel (albumin-bound) combined with oxaliplatin as the first-line drugs for treatment of advanced hepatobiliary and malignant tumors.

Primary endpoint: progression-free survival (PFS) Secondary study endpoints: disease control rate (DCR), overall survival (OS), and incidence and severity of adverse events (AE).

3 Research plan 3.1 Research Design This study was a single-center, one-arm, phase II/III clinical trial, which plans to recruit 57 patients.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients are ≥ 18 years old; 2) Pathological diagnosis confirmed advanced hepatocellular carcinoma, intrahepatic cholangiocellular carcinoma, extrahepatic cholangiocellular carcinoma, gallbladder carcinoma and pancreatic cancer by histopathological examination; 3) Having at least one measurable lesion according to the RECIST 1.1 tumor evaluation criteria; 4) Estimated survival time > 3 months; 5) There are no other concurrent anti-cancer treatments (including local radiotherapy and molecular targeted therapy, etc.) or previous treatment history; 6) ECOG PS score ≤ 2 points; 7) Cardiac color Doppler examination indicates a left ventricular ejection fraction (LVEF) ≥ 50%; 8) Having no obvious signs of hematological disease, ANC≥1.5×109/L, platelet count≥100×109/L, Hb≥90g/L, WBC≥3.0×109/L, and no bleeding tendency before enrollment; 9) Liver function test: total bilirubin (TBIL) is ≤ 1.5 times the upper limit of normal value, alanine aminotransferase (ALT), aspartate aminotransferase (AST) are ≤ 2.5 times the upper limit of normal value; renal function test: serum creatinine (Cr) ≤ 1.5mg/dl, or calculated creatinine clearance ≥50ml/min; 10) Patients can understand and sign the informed consent form.

Exclusion Criteria:

* 1) Pregnant or lactating female patients (women of childbearing age must be confirmed to have negative pregnancy test results within 7 days prior to the first dose, if they are positive, ultrasound examination is required to be performed to exclude pregnancy); women of childbearing age refuse to receive contraception.

  2) Having other malignant tumors, except cured basal cell carcinoma of the skin or squamous cell carcinoma of the skin or in situ carcinoma in any other regions; 3) Having abnormal bone marrow hyperplasia and other hematopoietic disorders; 4) Having active infections, HIV infection, and viral hepatitis that require systemic treatment; 5) Child-Pugh score > 7 points; 6) Being combined with medium-large ascites or hepatic encephalopathy; 7) Subjects with ≥1 peripheral neuropathy according to the National Cancer Institute Common Toxicity Response Standard (NCI-CTC) version 5.0; 8)Patients with severe cardiovascular diseases such as cerebrovascular accidents occurring within 6 months, myocardial infarction, hypertension that cannot be controlled after drug intervention, unstable angina pectoris, heart failure (NYHA 2-4), and arrhythmia requiring drugs intervention; 9) Being allergic to the drug or drug ingredients used in this test or having hypersensitivity history; 10) Having received any other drug treatment or participated in another interventional clinical trial within 30 days of the screening period; 11) Having dementia, mental state changes or any mental illness that may interfere with understanding or making informed consent or completing a questionnaire; 12) Being considered to be unsuitable for enrollment by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2019-08-20 (Estimated); Primary Completion 2021-04-20 (Estimated); Study Completion 2023-10-20 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 years
  Progression-free surviva

SECONDARY OUTCOMES:
DCR | 2 years
  Disease control rate
OS | 2 years
  overall survival
AE | 2 years
  incidence and severity of adverse events